#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for a phase I open-label, dose escalation study to investigate the safety, pharmacokinetics pharmacodynamics and clinical activity of GSK2879552 given orally in subjects with relapsed/refractory acute myeloid leukemia |
|---|---|---|
| <b>Compound Number</b> | : | GSK2879552 |
| <b>Effective Date</b> | : | 26-JUN-2018 |

#### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 2013N163643\_05.
- This RAP is intended to describe the safety, efficacy and pharmacokinetic analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Part 1 Statistical Analysis Complete (SAC) deliverable. Due to early termination of the study, Part 2 was not initiated. This document will only include the reporting plan for subjects enrolled in the study.

#### **RAP Author(s):**

| Authors: | Date | Approval Method |
|------------------------------------------|------|-----------------|
| PPD | NI A | NI A |
| Lead Statistician (Oncology, SPDS-India) | N. A | N. A |

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

## The GlaxoSmithKline group of companies

## **RAP Team Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Clinical Development (Oncology, ES Clinical) | 26-JUN-2018 | Email |
| Clinical Development Manager (Oncology CPSSO) | 21-JUN-2018 | Email |
| Director (Clinical Pharmacology, Modelling and Simulation) | 21-JUN-2018 | Email |
| Associate Manager (Oncology, SPDS-India) | 26-JUN-2018 | Email |
| Statistics Leader, (Oncology, Clinical Statistics) | 25-JUN-2018 | Email |
| Data Quality Lead | 24-JUN-2018 | Email |

## **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| General Manager, Biostatistics and Programming (Oncology, SPDS-India) | 26-JUN-2018 | Email |
| Biostatistics and Programming Manager (Oncology, SPDS-India) | 26-JUN-2018 | Email |

## **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTRODU | CTION | 5 |
| 2. | 2.1. Ch | Y OF KEY PROTOCOL INFORMATIONanges to the Protocol Defined Statistical Analysis Plan | 6 |
| | | udy Designatistical Analyses | |
| 3. | 3.1. Inte | ANALYSESerim Analyses | 12 |
| | | al Analyses | |
| 4. | | S POPULATIONSotocol Deviations | |
| 5. | | RATIONS FOR DATA ANALYSES AND DATA HANDLING | |
| | | TIONS | |
| | | udy Treatment & Sub-group Display Descriptorsseline Definitions | |
| | 5.3. Oth | ner Considerations for Data Analyses and Data Handling nventions | |
| 6. | STUDY PO | OPULATION ANALYSES | 16 |
| | | erview of Planned Study Population Analyses | |
| | | sposition of Subjectsbtocol Deviations | |
| | | mographic and Baseline Characteristics | |
| | | ncomitant Medications | |
| | | tent of Exposure | |
| 7. | | NALYSES | |
| | | verse Events Analyses | |
| | | verse Events of Special Interestnical Laboratory Analyses | |
| | 7.3. CIII<br>7.3 | | |
| | _ | ner Safety Analyses | |
| 8. | EFFICACY | Y ANALYSES | 23 |
| 9. | | COKINETIC ANALYSES | |
| | | mary Pharmacokinetic Analyses | |
| | 9.1 | The second secon | |
| | | 9.1.1.1. Drug Concentration Measures | |
| | 9.1 | | |
| | 9.1 | • | |
| | | 9.1.3.1. Dose proportionality | 25 |
| | | 9.1.3.2 Accumulation | 26 |

#### CONFIDENTIAL

| | | | 9.1.3.3. | Time Invariance | 26 |
|---|---|---|---|---|---|
| 10. | REFE | RENCES. | | | 27 |
| 11 | A DDE | UDICES | | | 20 |
| 11. | 11.1. | | | ol Deviation Management and Definitions for Per | 20 |
| | 11.1. | | | | 28 |
| | | | | s from Per Protocol Population | |
| | 11.2. | | | ule of Activities | |
| | 11.2. | 11 2 1 | Protocol D | Defined Schedule of Events | 29 |
| | 11.3. | | | ment Windows | |
| | 11.4. | | | Phases and Treatment Emergent Adverse | |
| | | Events | t i. Clady i | | 31 |
| | | | | ises | |
| | | | | Study Phases for Concomitant Medication | |
| | 11.5. | Appendix | | isplay Standards & Handling Conventions | |
| | | 11.5.1. | Reporting | Process | 32 |
| | | 11.5.2. | | Standards | |
| | | 11.5.3. | | Standards for Pharmacokinetic | |
| | 11.6. | Appendix | | d and Transformed Data | |
| | | 11.6.1. | General | | 34 |
| | | 11.6.2. | Study Pop | pulation | 34 |
| | 11.7. | Appendix | x 7: Reporti | ing Standards for Missing Data | 35 |
| | | 11.7.1. | | · Withdrawals | |
| | | 11.7.2. | | of Missing Data | |
| | | | | Handling of Missing and Partial Dates | |
| | | 11.7.3. | Imputation | n of Missing Exposure End Dates | 38 |
| | 11.8. | | | of Potential Clinical Importance | |
| | | | | y Values | |
| | 11.9. | | | iations & Trade Marks | |
| | | 11.9.1. | | ons | |
| | | 11.9.2. | | ks | |
| | 11.10. | | | Data Displays | |
| | | | • | lay Numbering | |
| | | | | mple Shell Referencing | |
| | | | | es | |
| | | | | oulation Tables | |
| | | | | ables | |
| | | 11.10.6. | Satety Tal | bles | 46 |
| | | | | kinetic Tables | |
| | | | | gs | |
| | 44.44 | | | _istings | |
| | 11.11. | Appendix | x 11: | ple Mock Shells for Data Displays | 56 |

#### 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol:

| GlaxoSmithKline<br>Document<br>Number | Date | Version |
|---------------------------------------|-------------|------------------|
| 2013N163643_00 | 2014-MAY-02 | Original |
| 2013N163643_01 | 2014-OCT-01 | Amendment No. 01 |

DLT criteria are revised according to the regulatory agency request. PD sampling requirements and subject populations are also clarified.

| 2013N163643_02 | 2015-MAY-27 | Amendment No. 02 |
|----------------|-------------|------------------|

Additional eligibility criteria and safety monitoring measures are put in place to address recent safety findings.

| 2013N163643_03 | 2016-MAY-09 | Amendment No.03 |
|----------------|-------------|-----------------|
|----------------|-------------|-----------------|

A combination arm with ATRA is added. One of the Dose Limiting Toxicities criteria has been revised according to the NCI criteria. Pharmacodynamic/exploratory sample collection and processing have been changed. Pharmacogenetic sample has been added. The criteria for Progressive Disease and Stable Disease have been added in the response criteria. Concomitant medications have been updated.

| 2013N163643_04 | 2017-MAY-02 | Amendment No. 4 |
|----------------|-------------|-----------------|
|----------------|-------------|-----------------|

Add language to include a stopping rule that halts enrollment upon the occurrence of any encephalopathy, unless clearly attributable to central nervous system disease involvement or intercurrent illness.

| 2013N163643_05 | 2017-OCT-06 | Amendment No. 5 |
|----------------|-------------|-----------------|
|----------------|-------------|-----------------|

Modify renal entrance criteria to align with regulatory agencies. Add additional dose adjustment language for hematologic toxicities. Optimize DLT criteria and safety management for retinoic acid syndrome. Add de-escalation language for both GSK2879552 and ATRA. Move PD secondary objective and endpoint to exploratory. Clarified definition of objective response rate (ORR). Included duration of response (DoR), time to response (TTR) and progression-free survival (PFS) as the secondary objectives in the expansion cohort. Updated statistical section to clarify data from Part 1 and Part 2 may be combined for analyses if appropriate. Deleted "dose limiting toxicity" as the safety endpoint of expansion cohort. Update and clarify inconsistencies within protocol: update dose escalation committee language to align with new standard language, define the "baseline" MOCA, baseline assessment of vitamin B12, TSH, free T3 or free T4 added at screening visit, define time window for informed consent, clarify urine metabolite and PK sample collections, add morphology to analysis of bone marrow

aspirates, clarify use of azoles permitted on study and other administrative updates.

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

## 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Due to the early termination of the study 200200, this RAP is developed for an abbreviated CPSR. Since Part 2 cohort expansion was not initiated prior to study closure, no statistical analysis will be performed for Part 2.

Changes from the originally planned statistical analysis specified in the protocol are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| Interim Analysis and CSR for<br>Part 2 | No Statistical Analysis for<br>Part 2 | Part 2 was not implemented |
| Full CSR | Abbreviated CSR | Study terminated |
| Pharmacokinetic Analysis of<br>ATRA for Part 1 | Pharmacokinetic Analysis of ATRA for Part 1 will not be performed | ATRA samples not provided to the analytical lab with adequate protection to light resulting in a very limited number of analysable samples which concentration are listed. |

## 2.2. Study Objective(s) and Endpoint(s)

| Part 1 Objectives | Part 1 Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To determine the safety, tolerability,<br>MTD and/or RP2D and regimen of<br>GSK2879552, alone or in combination<br>with ATRA, given orally in adult<br>subjects with AML. | AEs, SAEs, dose limiting toxicities, dose reductions or delays, withdrawals due to toxicities and changes in safety parameters (e.g., laboratory values, vital signs, electrocardiograms [ECGs], physical examinations). |
| Secondary Objectives | Secondary Endpoints |
| To characterize the PK of<br>GSK2879552, alone or in<br>combination with ATRA, after<br>single and repeat-dose oral<br>administration. | <ul> <li>GSK2879552 PK parameters following single-(Day 1) and<br/>repeat-dose (Day 15) administration of GSK2879552,<br/>including AUC, Cmax, tmax, t½ (terminal phase and/or<br/>effective half-life), accumulation ratio, and time invariance</li> </ul> |
| To evaluate clinical response after<br>treatment with GSK2879552, alone or<br>in combination with ATRA. | Objective response rate defined as the percentage of subjects achieving complete remission (CR), partial remission (PR), CRp (as per CR but platelet). |

| Part 1 Objectives | Part 1 Endpoints |
|---|---|
| • | Count <100 x 109/L) and morphologic leukemia free state per response criteria (Cheson, 2003). |
| To characterize the PK of ATRA in<br>combination with GSK2879552 after<br>single and repeat-dose oral<br>administration. | ATRA PK parameters following single and repeat-dose administration of ATRA and GSK2879552, including AUC, Cmax, tmax, t½ (terminal phase) . |
| Exploratory Objectives | Exploratory Endpoints |
| To explore markers of differentiation<br>(including morphology) in response to<br>GSK2879552, alone or in<br>combination with ATRA. | Change from baseline expression in cell surface markers in AML cells derived from bone marrow and/or peripheral blood. |
| To investigate the mechanism of action and indicators of sensitivity and resistance to GSK2879552, alone or in combination with ATRA. | Analysis of morphology, DNA, RNA and/or protein markers in blasts cells in bone marrow aspirates and/or peripheral blood. |
| To evaluate the relationship between<br>GSK2879552 exposure, alone or in<br>combination with ATRA and<br>safety/efficacy/PD parameters. | Relationship between GSK2879552 exposure markers (e.g. dose, concentration, Cmax, Cmin or AUC (0-tau)) and safety/efficacy/PD parameters. PD parameters assessed by change from baseline in select biomarkers, e.g. CD86 and CD11b |
| To characterize the metabolite profile<br>of GSK2879552 after oral single and<br>repeat-dosing in some subjects | GSK2879552 metabolites in plasma<br>and/or urine |
| To determine the amount of<br>GSK2879552 excreted in urine after<br>oral single and repeat dosing in some<br>subjects treated with GSK2879552 | Concentration of GSK2879552 in urine<br>measured with an investigational bioanalytical<br>method and extrapolated to total amount excreted in urine<br>over time. |
| To investigate the relationship<br>between genetic variants in candidate<br>genes, PK and safety profile of<br>GSK2879552, alone or in<br>combination with ATRA. | Pharmacogenomic (PGx) study using buccal samples. |

| Part 2 Objectives | Part 2 Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To evaluate clinical activity of<br>GSK2879552, alone or in<br>combination with ATRA at the<br>respective RP2D given orally in<br>adult subjects with AML. | Objective response rate defined as the percentage of subjects achieving complete remission (CR), partial remission (PR), CRp (as per CR but platelet Count <100 x 109/L) and morphologic leukemia free state per response criteria (Cheson, 2003). |
| Secondary Objectives | Secondary Endpoints |
| To evaluate the safety and<br>tolerability of respective RP2D of<br>GSK2879552, alone or in | AEs, SAEs, dose reductions or delays, withdrawals due to toxicities and changes in safety assessments (e.g., laboratory parameters, vital signs, ECGs, physical |

| Part 2 Objectives | Part 2 Endpoints |
|---|---|
| combination with ATRA. | examinations). |
| To characterize the population PK of<br>GSK2879552, alone or in combination<br>with ATRA. | <ul> <li>Population PK parameters for GSK2879552 such as<br/>clearance (CL/F) and volume of distribution (V/F), and<br/>relevant covariates which may influence<br/>exposure (e.g., age, weight, or disease<br/>associated covariates).</li> </ul> |
| To evaluate clinical activity in terms of duration of response, time to response (TTR) and progression free survival (PFS) | <ul> <li>Duration of response (DoR), defined as the time from first documented evidence of PR or better until disease progression (PD) or death, among responders, i.e. confirmed PR or better.</li> <li>Time to Response is defined as the time from first dose to the first documented evidence of response (PR or better).</li> <li>Progression-free survival (PFS), defined as the time from first dose until the earliest date of disease progression (PD), or death due to any cause.</li> </ul> |
| Exploratory Objectives | Exploratory Endpoints |
| To investigate the mechanism of action and indicators of sensitivity and resistance to GSK2879552, alone or in combination with ATRA. | <ul> <li>Analysis of morphology, DNA, RNA<br/>and/or protein markers in blast cells from bone marrow<br/>aspirate and/or peripheral blood sample.</li> </ul> |
| To evaluate the exposure response<br>(PK/PD) relationship between<br>GSK2879552, alone or in<br>combination with ATRA and<br>safety/efficacy/PD parameters. | Relationship between GSK2879552 exposure markers (e.g. dose, concentration, Cmax or AUC (0-tau)) and safety/efficacy/PD parameters. PD parameters assessed by change from baseline in select biomarkers, e.g. CD86 and CD11b |
| To investigate the relationship<br>between genetic variants in<br>candidate genes, PK and safety<br>profile of GSK2879552, alone or in<br>combination with ATRA. | Pharmacogenomic (PGx) study using buccal samples |

#### 2.3. Study Design



- PK/PD expansion: Any dose level could be expanded up to 12 subjects during dose escalation.
- Alternative dosing schedule may be explored.

## Design Features

Part 1: Dose Escalation Phase

#### GSK2879552 Monotherapy

- In Cohort 1, a single subject will receive a dose of GSK2879552 1 mg once daily. The subject in Cohort 1will be evaluated for dose limiting toxicities (DLTs) during the first 4 weeks of treatment (DLT observation window), and the safety and PK data will be reviewed prior to a dose escalation decision and starting Cohort 2. If the first subject becomes unevaluable for reasons other than toxicity, another subject will be recruited. The dose-escalation decision and rationale will be documented in writing with copies maintained at each study site and in the master study files at GlaxoSmithKline (GSK).
- Starting with Cohort 2, the dose escalation will continue using the Neuenschwander continuous reassessment method (N-CRM) [Neuenschwander, 2008]. A sufficient
  number of subjects will be enrolled in each cohort to ensure that data from at least
  one subject that has completed the DLT observation window is available prior to
  defining a new dose and starting the next cohort. In addition, subjects who fail to take
  at least 75% of their scheduled doses in the 4 weeks for reasons other than toxicity
  will be replaced.

#### GSK2879552 and ATRA combination

In Cohort 1, three subjects will receive GSK2879552 2 mg once daily. After all three subjects complete the first 4 weeks of treatment, the safety data will be reviewed for DLT. Available PK and PD data will be also reviewed prior to a dose escalation decision and starting Cohort 2. Each cohort will enroll 3 or more subjects to obtain sufficient data. If any subject becomes unevaluable for reasons other than toxicity, a replacement subject will be enrolled. In addition, subjects who fail to take at least 75%

### **Overview of Study Design and Key Features** of their scheduled doses of each drug in the first 4 weeks for reasons other than toxicity will be replaced. Starting with Cohort1, the dose escalation will use the N-CRM with prior DLT information of GSK2879552 and ATRA monotherapies and follow the same rule with regards to the number of subjects, maximum dose increment, and the completion of dose escalation as in Monotherapy. PK/PD Expansion Cohort Any dose level(s) in Part 1 may be expanded up to 12 subjects in order to collect adequate data on safety. PK or PD. However, PD sample (peripheral blood and bone marrow aspirate) collection may be stopped early at the sponsor's discretion. Subjects may be enrolled at previously completed dose levels for the purpose of obtaining additional data. These subjects may have the dose escalated to a higher completed dose level (not exceeding the maximum tolerated dose [MTD]) once the necessary PK/PD procedures have been completed. Part 2: Expansion Cohort Once the respective RP2D have been determined, an expansion cohort of up to 30 subjects each, GSK2879552 mono-therapy or in combination with ATRA, will be enrolled in order to better characterize the clinical activity and safety profile of the RP2D. Additional expansion cohorts may be initiated to test the efficacy of i) GSK2879552 at RP2D in ≥60 years old treatment naïve subjects, and ii) GSK2879552 in combination with other agents (demonstrated synergy in pre-clinical studies) in relapsed/refractory or ≥60 years old treatment naïve subjects. The statistical design and number of subjects to be enrolled in the dose expansion cohort is based on the predictive probability of success if enrollment continues until all planned subjects are recruited [Lee, 2008]. The predictive probability design allows for evaluation of stopping rules after each subject once a minimum number of subjects are evaluable. In this particular study, we will stop only for futility. Futility analysis for each dose expansion cohort will begin when response data is available for at least 10 evaluable subjects. The dose expansion cohort may be stopped early for futility if the predictive probability of success (response rate ≥ historical response rate) is less than 5%. Dosing In Part 1, in Cohort 1, a single subject will receive a dose of GSK2879552 1 mg once daily. The subject in Cohort 1 must complete a full 28 days of dosing, and the safety and PK data will be reviewed prior to starting Cohort 2. Starting with Cohort 2 the dose escalation will continue using the Neuenschwander continuous reassessment method (N-CRM). Upon review of the safety, tolerability, clinical activity, PK, PD data, the RP2D or doses will be selected. Subjects may be enrolled at previously completed dose levels for the purpose of obtaining additional PK or PD data. In Part 2, once the RP2D has been determined, subjects will be enrolled at the RP2D and will be evaluated for safety and efficacy while monitoring the futility stopping rules. Time & Refer to Protocol Amendment 5 Section 7.1 Time and Event Table(s)

**Events** 

| Overview of St | udy Design and Key Features |
|---|---|
| Treatment | Subjects will be identified by a unique subject number that will remain consistent for the |
| Assignment | duration of the study, except for subjects who are allowed intra-subject dose escalation |
| | and start the treatment from Day 1 with the new subject numbers allocated to them. |
| Interim<br>Analysis | <ul> <li>In Part 1, interim analyses to inform dose escalation will be performed following the completion of each monotherapy and combination dose cohort in part 1. The primary driver for dose escalation decisions in Part 1 will be governed by an N-CRM model for the mono-therapy dose cohorts and a Bayesian copula regression for the combination dose cohorts. They will be used to predict the probability of DLT at the dose levels yet to be tested to further guide these decisions.</li> <li>After the initial 10 evaluable subjects, have enrolled at the RP2D dose, response data will be reviewed on an ongoing basis and the number of responses observed will be compared with the stopping rules provided in Section 13.4.2 of Protocol Amendment 5.</li> </ul> |

#### NOTES:

 Due to the business decision of study termination, Part 2 was not implemented. As a result, the remainder of this document contains no content related to Part 2 and will only provide information related to Part 1.

## 2.4. Statistical Hypotheses / Statistical Analyses

No formal statistical hypotheses are being tested. Analysis of the data obtained from this study will be focused on comparison between dose cohorts and only descriptive methods will be used in analysis of the data obtained from this study.

#### 3. PLANNED ANALYSES

### 3.1. Interim Analyses

In Part 1, interim analyses to inform dose escalation will be performed following the completion of each monotherapy and combination dose cohort in part 1. The primary driver for dose escalation decisions in Part 1 will be governed by a N-CRM model for the mono-therapy dose cohorts and a Bayesian copula regression for the combination dose cohorts. They will be used to predict the probability of DLT at the dose levels yet to be tested to further guide these decisions.

Interim analysis on Part 1 may also be conducted when all subjects enrolled in Part 1 have had at least one post-baseline disease assessments or progressed or died or withdrawn from the study.

Additionally, safety, PK, PD/biomarker data may be examined during Part 1. Prior to determining GSK2879552 dose for the next monotherapy cohort, exploratory analysis maybe conducted to assess the relationship of GSK2879552 dose levels with safety, PK and PD parameters using all data from available cohorts.

### 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.
- 2. All criteria for unblinding the randomization codes have been met.

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | All subjects who were screened for eligibility | Screen Failure |
| Enrolled | All participants who passed screening and entered the study. | <ul> <li>Number of participants by Country and Siteid</li> <li>Age Ranges</li> </ul> |
| All Treated<br>Subjects | All randomized participants who received at least one dose of study treatment. | Study Pop, Safety,<br>Efficacy |
| Pharmacokinetic | All treated subjects for whom a PK sample is obtained and analysed. | • PK |
| Pharmacodynamic | All treated subjects who contribute to PD/Biomarker samples. | • PD |

Refer to Appendix 10 List of Data Displays which details the population used for each display.

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.

Data will be reviewed prior to freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.

o This dataset will be the basis for the listings of protocol deviations.

A separate listing of all inclusion/exclusion criteria deviations will also be provided.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

## 5.1. Study Treatment & Sub-group Display Descriptors

| | | Data Displays for Reporting | |
|------|-------------|-----------------------------|--------------|
| Code | Description | Description | Order in TLF |
| Α | GSK2879552 | 1mg QD | 1 |
| | | 2mg QD | 2 |
| | | 4mg QD | 3 |
| | | 8mg QD | 4 |
| | | 12mg QD | 5 |
| | | 20mg QD | 6 |
| | | 2mg QD/ATRA<br>45mg/m2/day | 7 |
| | | 20mg QD PK/PD<br>EXPANSION | 8 |

## 5.2. Baseline Definitions

• Baseline will be defined as the most recent, non-missing value prior to or on the first study treatment dose date.

# 5.3. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 11.3 | Appendix 3: Assessment Windows |
| 11.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 11.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 11.5 | Appendix 6: Derived and Transformed Data |
| 11.7 | Appendix 7: Reporting Standards for Missing Data |
| 11.8 | Appendix 8: Values of Potential Clinical Importance |

#### 6. STUDY POPULATION ANALYSES

#### 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the All Treated Subjects population, unless otherwise specified.

Study population analyses will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 10: List of Data Displays.

### 6.2. Disposition of Subjects

A summary of subject status and reason for study withdrawal will be provided. This display will show the number and percentage of subjects who withdrew from the study, including primary reasons for study withdrawal. Reasons for study withdrawal will be presented in the order they are displayed in the eCRF. A listing of reasons for treatment discontinuation will also be provided. A listing of reasons for screen failure will also be provided.

#### 6.3. Protocol Deviations

Important protocol deviations will be listed and will include inclusion and exclusion deviations as well as other deviations.

Participants excluded from any population will be listed.

## 6.4. Demographic and Baseline Characteristics

The demographic characteristics (e.g., age, race, ethnicity, sex, baseline height, and baseline body weight will be summarized and listed. Age, height and weight will be summarized using the mean, standard deviation, minimum, median, and maximum. In addition, age will also be categorized and summarized by 18-64, >=65-84, and >=85. The count and percentage will be computed for sex and ethnicity. A separate summary of age ranges will be produced for study disclosure requirements.

Race and racial combinations will be summarized. A listing of race will also be provided.

Current and past medical conditions will be summarized and listed.

Prior anti-cancer therapy will be coded using GSK Drug coding dictionary. A listing of prior anti-cancer therapy will show ATC Level 1, Ingredient, and verbatim text. Prior anti-cancer therapy and prior cancer related surgeries will be listed.

Disease Characteristics at Screening will be listed.

A listing of substance use will also be provided.

#### 6.5. Concomitant Medications

Concomitant medications will be coded using GSK Drug coding dictionary and summarized. The summary of concomitant medications will show the number and percentage of subjects taking concomitant medications by Ingredient. Concomitant Medications will be listed.

#### 6.6. Extent of Exposure

Extent of exposure of GSK2879552, alone or in combination with ATRA will depend on tolerability of the subjects to the doses administered and the course of their disease. The number of subjects exposed to GSK2879552, alone or in combination with ATRA will be summarized for each dose level administered according to the duration of therapy. The duration of exposure to study treatment in weeks (from first day to last day of treatment plus) will also be summarised.

All the dose reductions, dose escalations and dose interruptions will be summarised and listed separately.

.

#### 7. SAFETY ANALYSES

The safety analyses will be based on the All Treated Subjects population, unless otherwise specified. All summaries will be presented by dose level.

Study population analyses will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 10: List of Data Displays.

#### 7.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), serious AEs (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 10: List of Data Displays.

AEs will be graded according to the CTCAE, Version 4.0. Adverse events will be coded to the PT level using the MedDRA dictionary. The relationship of AE system organ, preferred term, and verbatim text will be listed. The subject numbers for individual AEs will be listed.

A summary of number and percentage of subjects with any adverse events by maximum grade will be produced. AEs will be sorted by System Organ Class (SOC) and Preferred term (PT) in descending order of total incidence.

The relationship between MedDRA SOC, PT, and Verbatim Text will be listed.

A listing of All AEs will be provided.

Serious adverse events by system organ class and preferred term (number of participants and occurrences) will be summarized. All serious adverse events (SAEs) will be tabulated based on the number and percentage of subjects who experienced the event. The summary tables will be displayed in descending order of total incidence.

Separate listings will be generated for all fatal SAEs and non-fatal SAEs.

## 7.2. Adverse Events of Special Interest

A comprehensive list of MedDRA terms based on clinical review will be used to identify each of the AESI.

The events of special interest include:

- Encepalopathy
- Thrombocytopenia
- Hemorrhages
- Diarrhea

- Nausea & Vomiting
- Constipation
- Infections
- Neutropenia
- Fatigue
- Anemia

One summary giving number and percentage of subjects for each of these AESI will be provided. Separate listing for each of the AESI will also be provided.

## 7.3. Clinical Laboratory Analyses

Laboratory evaluations will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 10: List of Data Displays.

The assessment of laboratory toxicities will examine the following laboratory tests as specified in Table 2 below.

Table 2 Laboratory Tests

| Hematology |
|---|
| Platelet count |
| White blood cell (WBC) Count (absolute) |
| Hemoglobin |
| Automated WBC Differential: |
| Neutrophils |
| Lymphocytes |
| Monocytes |
| Eosinophils |
| Basophils |
| Red blood cell (RBC) Indices (at screening and if Hemoglobin decrease ≥2 g/dL compared to baseline): |
| Mean corpuscular volume (MCV) |
| Mean corpuscular hemoglobin( MCH) |
| Mean corpuscular hemoglobin concentration (MCHC) |
| Reticulocytes |
| RBC |

| Clinical Chemistry | | | |
|---|---|---|---|
| Blood urea | Potassium | Aspartate aminotransferase (AST) | Total and Direct bilirubin1 |
| nitrogen | | | |
| Creatinine | Chloride | Alanine aminotransferase (ALT) | |
| Glucose, random | Total CO2 | Albumin | |
| Sodium | Calcium <sup>2</sup> | Alkaline phosphatase (ALP) | |
| Magnesium | Phosphorus | Lactate dehydrogenase (LDH) | |
| Fasting Lipid panel i | including fraction | ated serum cholesterol, triglycerides, tota | al cholesterol, HDL and LDL |
| Estimated glomerula | ar filtration (Modit | ication of Diet in Renal Disease) or 24 hr | urine creatinine clearance <sup>3</sup> |
| Beta-hCG pregnand | y test for approp | riate females (serum or urine) | |
| Coagulation | | | |
| Prothrombin time/International normalized ratio (PT/INR) | | | |
| Partial prothrombin time (PTT) | | | |
| Urinalysis | | | |
| Specific gravity | | | |
| pH – dipstick | | | |
| Glucose – dipstick | | | |
| Protein – dipstick | | | |
| Blood – dipstick | | | |
| Ketones – dipstick | | | |
| Microscopic examination required (if blood or protein by dipstick ≥1+) | | | |
| Urine total protein to creatinine ratio (UPC ratio) – (if protein by dipstick ≥2+) | | | |

- 1. Bilirubin fractionation is required if total bilirubin >2x ULN
- 2. For screening ionized calcium is acceptable
- The Modification of Diet in Renal Disease Equation will be used to determine an estimated glomerular filtration rate.

Laboratory grades will be reported using the Common Terminology Criteria for Adverse Events (CTCAE v4.0).

For hematology, RBC is not gradable by CTCAE v4.0.

For clinical chemistry, BUN, LDH and estimated creatinine clearance are not gradable by CTCAE v4.0.

For coagulation tests, INR and partial thromboplastin time are gradable by CTCAE v4.0 but prothrombin time is not.

For all laboratory results, displays for hematology, clinical chemistry, and liver function tests will be separately produced.

Summaries of worst case grade increase from baseline grade will be provided for all the lab tests that are gradable by CTCAE v4.0. These summaries will display the number and percentage of subjects with a maximum post-baseline grade increasing from their baseline grade. Any increase in grade from baseline will be summarized along with any increase to a maximum grade of 3 and any increase to a maximum grade of 4. Missing baseline grade will be assumed as grade 0. For laboratory tests that are graded for both

low and high values, summaries will be done separately and labeled by direction, e.g., sodium will be summarized as hyponatremia and hypernatremia.

For lab tests that are not gradable by CTCAE v4.0, summaries of worst case changes from baseline with respect to normal range will be generated. Decreases to low, changes to normal or no changes from baseline, and increases to high will be summarized for the worst case post-baseline. If a subject has a decrease to low and an increase to high during the post-baseline time period, then the subject is counted in both the "Decrease to Low" categories and the "Increase to High" categories.

A supporting listing of all chemistry and haematology laboratory data will be provided.

Unless otherwise specified, the denominator in percentage calculation at each scheduled visit will be based on the number of subjects with non-missing value at each particular visit.

#### 7.3.1. Liver Function Analyses

Summaries of hepatobiliary laboratory events including possible Hy's law cases will be provided in addition to what has been described above.

Possible Hy's law cases are defined as any elevated (ALT>3×ULN **and** total bilirubin  $\ge 2 \times \text{ULN}$  (with direct bilirubin  $\ge 35\%$  of total bilirubin, if direct bilirubin is measured)) **OR** (ALT  $\ge 3$  times ULN **and** INR >1.5, if INR is measured).

### 7.4. Other Safety Analyses

The analyses of non-laboratory safety assessment results will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 10: List of Data Displays.

Unless otherwise specified, the denominator in percentage calculation at each scheduled visit will be based on the number of subjects with non-missing value at each particular visit.

#### **ECG**

A summary of the number and percentage of subjects who had normal and abnormal (clinically significant and not clinically significant) ECG findings will be displayed by scheduled visits as well as for the worst case post-baseline. The summaries for the QTc will use the collected value based on QTcB and QTcF.

The QTcB and QTcF values will be rounded to the integer and the values will be categorized into the following ranges: Grade 0 (<450), Grade 1 (450-480), Grade 2 (481-500), and Grade 3 (≥501). Summaries of grades will display the number and percentage of subjects by grade in the worst case post-baseline. Similarly, grade changes relative to baseline grade will also be generated.

Listings of abnormal ECG findings and a listing of ECG values will be provided.

#### Vital Signs

Changes in heart rate from baseline, Increase in Blood Pressure from baseline and changes in Temperature from baseline will be summarised.

A separate listing of vital signs will also be produced.

#### **Left Ventricular Ejection Fraction**

A listing of the left ventricular ejection fraction results will be generated.

#### **ECOG Performance Status**

A summary of change from baseline in ECOG performance status by scheduled visits will be performed. Summaries will use frequency and percentage of subjects at each planned assessment time, best and worst-case post baseline.

A supporting listing will also be provided.

#### **Montreal Cognitive Assessment (MOCA)**

A listing of the Montreal Cognitive Assessment will be generated.

#### 8. EFFICACY ANALYSES

All efficacy analyses will be based on the All Treated Subjects population unless otherwise specified. All analyses will be presented by dose of study treatment. Details of the planned displays are provided in Appendix 10: List of Data Displays.

Response rate (RR) is defined as the percentage of subjects who achieved CR, CRp, PR or morphologic leukemia-free state (MLFS) among subjects who received at least one dose of treatment.

The investigator-assessed best response along with response rate (Without confirmation) will be summarized by dose of study treatment. A listing of investigator assessed responses (Without Confirmation) will be provided.

#### 9. PHARMACOKINETIC ANALYSES

#### 9.1. Primary Pharmacokinetic Analyses

Pharmacokinetic analysis will be the responsibility of the Clinical Pharmacology Modeling and Simulation (CPMS) Department, GSK.

The results of the pharmacokinetic analysis may be provided in a report separate from the main CSR.

#### 9.1.1. Endpoint / Variables

#### 9.1.1.1. Drug Concentration Measures

The GSK2879552 concentration-time data will be summarized by planned time point and dose cohort. Standard summary statistics will be calculated (i.e. mean, standard deviation, median, minimum and maximum). The ATRA concentration-time data will be listed.

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 11.5 Reporting Process & Standards).

#### 9.1.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic analysis of GSK2879552 will be conducted by noncompartmental methods using WinNonlin (Version 6.3 or higher). However pharmacokinetic analysis of ATRA will not be conducted due to the sample size limitations. The following pharmacokinetic parameters will be determined for if data permit:

| Parameter | Parameter Description |
|---|---|
| AUC(0-t) | Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (C(t)) will be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| AUC(0-τ) | Area under the concentration-time curve during a dosing interval of duration "tau". |
| AUC (0-∞) | Area under the concentration-time curve extrapolated to infinity will be calculated as: AUC = AUC(0-t) + C(t) / lambda_z |
| | This will be calculated for Day 1 only |
| Cmax | Maximum observed plasma concentration, determined directly from the concentration-time data. |
| tmax | Time to reach Cmax, determined directly from the concentration-time data. |
| t½ | Apparent terminal half-life will be calculated as: |
| | $t\frac{1}{2} = \ln 2 / \lambda z$ |
| λz | Apparent terminal phase elimination rate constant |
| Ст | Trough concentration |

To estimate the extent of accumulation after repeat dosing, the observed accumulation ratio (Ro) may be determined from the ratio of AUC(0- $\tau$ ) in Day 15/ AUC(0- $\tau$ ) in Day 1. The ratio of AUC(0- $\tau$ ) on Day 15/ Day 1 AUC(0- $\infty$ ) will be calculated to assess time invariance.

#### 9.1.2. Population of Interest

The primary pharmacokinetic analyses will be based on the Pharmacokinetic population, unless otherwise specified.

#### 9.1.3. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 9.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

Plasma concentration-time data for GSK2879552 and ATRA will be listed by dose and Plasma concentration-time data for GSK2879552 will be summarized using descriptive statistics (n, mean, standard deviation [SD], median, minimum and maximum) by planned relative assessment time. Mean and/ or median values will be plotted over time. Individual plasma and urinary (if available) PK parameters values as well as a descriptive summary (mean, standard deviation, median, minimum, maximum, geometric mean, and the standard deviation, Coefficient of variance [CV]% and 95% confidence interval of log-transformed parameters, if applicable) by dose cohort will be reported. The following pharmacokinetic statistical analyses will only be performed, if sufficient data is available.

#### 9.1.3.1. Dose proportionality

If data permits, dose proportionality will be assessed using power model for:

- AUC(0-∞) and Cmax on Day 1
- AUC(0- $\tau$ ) and Cmax on Day 15

Dose proportionality of GSK2879552 AUC(0- $\infty$ ) and Cmax following single dose administration and AUC(0- $\tau$ ) and Cmax following repeat dose administration will be evaluated using the power model as described below:

log (pharmacokinetic parameter) = a + b \* log(dose)

where a is the intercept and b is the slope.

The power model will be fitted by restricted maximum likelihood (REML) using SAS Proc Mixed. Both the intercept and slope will be fitted as fixed effects. If there is sufficient data, the model may also be fit with the intercept and/or slope as random effects depending on the ability of the model to converge and on estimation of variance-covariance matrix. The mean slope and corresponding 90% confidence interval will be estimated from the power model.

#### 9.1.3.2. Accumulation

If data permits, accumulation using ANOVA will be performed for AUC(0- $\tau$ ) on Day 15 vs AUC(0- $\tau$ ) on Day 1 by dose cohort.

To estimate the extent of accumulation after repeat dosing, the observed accumulation ratio (Ro) based on AUC data will be determined as follows:

$$Ro = AUC(0-\tau)_{D15}/AUC(0-\tau)_{D1}$$

Assuming both linear and time-invariant pharmacokinetics, the Ro at steady-state should be unity.

An ANOVA with a random effect term for subject and fixed effect terms for day will be performed by dose on the  $log_e$ -transformed PK parameters AUC(0- $\tau$ ). Day will be treated as a class variable in the model. The accumulation ratio of GSK2879552 will be estimated by calculating the ratio of the geometric least squares (GLS) means of the PK parameter between Day 15 and Day 1 for all dose levels and the corresponding 90% CI for each ratio.

The accumulation ratio will be summarized by dose.

#### 9.1.3.3. Time Invariance

To evaluate whether the pharmacokinetics remains unaltered after repeat dosing a similar analysis to that described above will be carried out after  $log_e$ -transformation of AUC(0- $\infty$ ) for D1 and AUC(0- $\tau$ ) for D15, the difference of which provides the steady-state ratio (Rs).

A mixed effect model will be fitted with day as a fixed effect and subject as a random effect for each treatment (dose) separately.  $AUC(0-\tau)$  on D15 will be compared to  $AUC(0-\infty)$  on D1 in order to assess time invariance for each dose. The Kenward & Roger (KR) degrees of freedom approach will be used. The ratio and 90% confidence interval will be calculated by back-transforming the difference between the least square means for the two days and associated 90% confidence interval, for each dose. Assuming both linear and time-invariant pharmacokinetics, the Rs at steady-state should be one.

The time invariance ratio will be summarized by dose.

#### 10. REFERENCES

Cheson BD et al. Revised recommendations of the International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia. J Clin Oncol. 2003; 21(24):4642-9.

GUI 137354 (2.0): Information for Authors: Reporting and Analysis Plans

GUI 51487: Non-compartmental Analysis of Pharmacokinetic Data, CPMS Global

Lee JJ, Liu DD. A predictive probability design for phase II cancer clinical trials. *Clinical Trials*. 2008; 5(2):93-106.

Neuenschwander B, Branson M, Gsponer T. Critical aspects of the Bayesian approach to phase I cancer trials, Stat in Med. 2008 27:2420-2439

SOP\_54838 (6.0): Development, Review and Approval of Reporting and Analysis Plans

## 11. APPENDICES

# 11.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

## 11.1.1. Exclusions from Per Protocol Population

There will be no Per Protocol population used for any displays or statistical analysis.

## 11.2. Appendix 2: Schedule of Activities

## 11.2.1. Protocol Defined Schedule of Events

Refer to Protocol Amendment 5 Section 7.1.

## 11.3. Appendix 3: Assessment Windows

No assessment windows will be applied.

## 11.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

## 11.4.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to treatment start date.

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Date < Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date ≤ Date ≤ Study Treatment Stop Date |
| Post-Treatment | nt Date > Study Treatment Stop Date |

#### 11.4.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is before 28 days prior to screening visit |
| Concomitant | Any medication that is not a prior |

#### NOTES:

 Please refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

## 11.5. Appendix 5: Data Display Standards & Handling Conventions

#### 11.5.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software will be used. | |
| Reporting Area | |
| HARP Server | : US1SALX00259 |
| HARP Compound | : Compound: GSK2879552, Study:200200 |
| Analysis Datasets | |
| Analysis datasets will be created according to Legacy GSK A&R dataset standards | |
| Generation of RTF Files | |
| RTF files will be generated for tables and figures. | |

#### 11.5.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### Planned and Actual Time

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days
    on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures, summaries and statistical analyses.

#### **Unscheduled Visits**

• Unscheduled visits will not be included in summary tables and figures.

| All unscheduled visits will be included in listings | |
|---|---|
| Descriptive Summary Statistics | |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

## 11.5.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Concentration Data | |
|---|---|
| PC Windows Non-<br>Linear (WNL) File | PC WNL file (CSV format) for the non-compartmental analysis by Clinical Pharmacology Modelling and Simulation function will be created according to [Insert document name]. Note: Concentration values will be imputed as per GUI_51487 |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1. Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. |
| Pharmacokinetic Parameter Data | |
| Is NQ impacted PK<br>Parameters Rule<br>Being Followed | Yes, refer to [Standards for Handling NQ Impacted PK Parameters]. |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to GUI_51487 |

#### 11.6. Appendix 6: Derived and Transformed Data

#### 11.6.1. General

#### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window the value closest to the target day for that window will be used. If values are the same distance from the target, then the mean will be taken.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### **Study Day**

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < First Dose Date → Study Day = Ref Date First Dose Date
  - Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

#### 11.6.2. Study Population

#### **Demography**

#### Age

- · Age will be calculated based on the Screening visit date
- Birth date will be imputed as follows:

Any subject with a missing day will have this imputed as day '15'.

Any subject with a missing date and month will have this imputed as '30JUN'.

#### **Body Mass Index**

Calculated as weight (kg) / [height (m)]2

#### **Extent of Exposure**

Number of days of exposure to study drug will be calculated based on the formula:

#### Duration of Exposure in Days = Treatment Stop Date - (Treatment Start Date) + 1

- Participants who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.
- The cumulative dose will be based on the formula:

#### **Cumulative Dose = Sum of (Number of Days x Total Daily Dose)**

- If there are any treatment breaks during the study, exposure data will be adjusted accordingly.
- Note: GSK2879552 exposure data will only be used for the above calculation.

#### 11.7. Appendix 7: Reporting Standards for Missing Data

#### 11.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>A subject will be considered to have completed the study if they complete screening<br/>assessments, at least 28 days of study treatment(s) and the post-treatment follow-up<br/>visit.</li> </ul> |
| | <ul> <li>If subjects which prematurely discontinue, additional subjects may be enrolled as<br/>replacement subjects at the discretion of the Sponsor in consultation with the<br/>investigator.</li> </ul> |
| | <ul> <li>Subjects who fail to take at least 75% of their scheduled doses in the first 28 days for<br/>reasons other than toxicity (e.g., dose limiting toxicities) will be replaced</li> </ul> |
| | <ul> <li>All available data from participants who were withdrawn from the study will be listed<br/>and all available planned data will be included in summary tables and figures, unless<br/>otherwise specified.</li> </ul> |
| | Withdrawal visits will be summarised as withdrawal visits. |

#### 11.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank field<br/>the collection instrument:</li> </ul> |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

#### 11.7.2.1. Handling of Missing and Partial Dates

Imputed partial dates will not be used to derive study day, duration (e.g. duration of adverse events), or elapsed time variables.

Imputed dates will not be displayed in listings. However, where necessary, display macros may impute dates as temporary variables for the purpose of sorting data in listings only. In addition, partial dates may be imputed for 'slotting' data to study time periods or for specific analysis purposes as outlined below.

| Dataset | Date | Missing | Rule |
|---|---|---|---|
| | | Element | |
| Adverse | Start | day, | <ul> <li>No Imputation for completely missing dates</li> </ul> |
| Events | Date | month, | |
| (AE) | | and year | |
| | | day, | • If study treatment start date is missing (i.e. subject did |

| Dataset | Date | Missing | Rule |
|---|---|---|---|
| Dutuset | Dutt | Element | |
| | | month | not start study treatment), then set start date = January 1. • Else if study treatment start date is not missing: o If year of start date = year of study treatment start date then • If stop date contains a full date and stop date is earlier than study treatment start date then set start date = January 1. • Else set start date = study treatment start date. o Else set start date = January 1. |
| | | Day | <ul> <li>If study treatment start date is missing (i.e. subject did not start study treatment), then set start date = 1st of month.</li> <li>Else if study treatment start date is not missing: <ul> <li>If month and year of start date = month and year of study treatment start date then</li> <li>If stop date contains a full date and stop date is earlier than study treatment start date then set start date= 1st of month.</li> <li>Else set start date = study treatment start date.</li> <li>Else set start date = 1st of month.</li> </ul> </li> </ul> |
| | End<br>Date | | No imputation for partial end dates will be performed |

## Concomitant Medication and Blood and Blood Supportive Care Products:

Start and end dates may be imputed for use in derivation of the reference variables concomitant medication start and end relative to treatment and blood and blood supportive care start and end relative to treatment, but should not be permanently stored in the analysis datasets.
| Dataset | Date | Missing<br>Element | Rule |
|---|---|---|---|
| Concomitant<br>Medication Blood and<br>Blood Supportive Care Products | Start<br>Date | day,<br>month,<br>and year | No Imputation for completely missing dates |
| | | day,<br>month | <ul> <li>If study treatment start date is missing (i.e. subject did not start study treatment), then set start date = January 1.</li> <li>Else if study treatment start date is not missing: <ul> <li>If year of start date = year of study treatment start date then</li> <li>If stop date contains a full date and stop date is earlier than study treatment start date then set start date = January 1.</li> <li>Else set start date = study treatment start date.</li> <li>Else set start date = January 1.</li> </ul> </li> </ul> |
| | | day | <ul> <li>If study treatment start date is missing (i.e. subject did not start study treatment), then set start date = 1st of month.</li> <li>Else if study treatment start date is not missing: <ul> <li>If month and year of start date = month and year of study treatment start date then</li> <li>If stop date contains a full date and stop date is earlier than study treatment start date then set start date= 1st of month.</li> <li>Else set start date = study treatment start date.</li> <li>Else set start date = 1st of month.</li> </ul> </li> </ul> |
| | End<br>Date | day,<br>month,<br>and year | No Imputation for completely missing dates |
| | | day,<br>month | • If partial end date contains year only, set end date = earliest of December 31 or date of last contact. |
| | | day | • If partial end date contains month and year, set end date = earliest of last day of the month or date of last contact. |

## 11.7.3. Imputation of Missing Exposure End Dates

For subjects who have missing end dates in their last exposure record potentially due to being lost to follow-up, the last contact date will be imputed as the last exposure date (i.e. date of last dose). This imputation will only be used when needed.

#### 11.8. Appendix 8: Values of Potential Clinical Importance

### 11.8.1. Laboratory Values

Reference ranges for all laboratory parameters collected throughout the study are provided by the laboratory. A laboratory value that is outside the reference range is considered either high abnormal (value above the upper limit of the reference range) or low abnormal (value below the lower limit of the reference range). Note: a high abnormal or low abnormal laboratory value is not necessarily of clinical concern. The laboratory reference ranges will be provided on the listings of laboratory data.

To identify laboratory values of potential clinical importance, National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE v4.0) will be used to assign grades to the relevant laboratory parameters.

# 11.9. Appendix 9: Abbreviations & Trade Marks

## 11.9.1. Abbreviations

| Abbreviation | Description |
|---|---|
| AE | Adverse Event |
| AESI | |
| ATRA | Adverse Events of Special Interest All Trans-Retinoic Acid |
| A&R | Analysis and Reporting |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CRF | Case Report Form |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTCAE | Common Terminology Criteria for Adverse Events |
| CTR | Clinical Trial Register |
| DBF | Database Freeze |
| DBR | Database Release |
| DOB | Date of Birth |
| DLT | Dose Limiting Toxicity |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| GSK | GlaxoSmithKline |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDSL | Integrated Data Standards Library |
| IP | Investigational Product |
| MOCA | Montreal Cognitive Assessment |
| MTD | Maximum Tolerated Dose |
| NCI | National Cancer Institute |
| PCI | Potential Clinical Importance |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PD | Pharmacodynamic |
| PP | Per Protocol |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RP2D | Recommended Phase 2 Dose |
| SAC | Statistical Analysis Complete |
| SOP | Standard Operation Procedure |
| | · |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |

## 11.9.2. Trademarks

| Trademarks of the GlaxoSmithKline |
|-----------------------------------|
| Group of Companies |

NONE

Trademarks not owned by the GlaxoSmithKline Group of Companies

SAS

WinNonlin

## 11.10. Appendix 10: List of Data Displays

### 11.10.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-------------|---------|
| Study Population | 1.1 to 1.15 | N. A |
| Efficacy | 2.1 | N. A |
| Safety | 3.1 to 3.20 | N. A |
| Pharmacokinetic | 4.1 to 4.6 | N. A |
| Section | List | ings |
| ICH Listings | 1 to 34 | |
| Other Listings | 35 to | o 48 |

## 11.10.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 11: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------------------------|----------|----------|----------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |
| Population Pharmacokinetic (PopPK) | POPPK_Fn | POPPK_Tn | POPPK_Ln |
| Pharmacodynamic and / or Biomarker | PD_Fn | PD_Tn | PD_Ln |
| Pharmacokinetic / Pharmacodynamic | PKPD_Fn | PKPD_Tn | PK/PD_Ln |

#### NOTES:

#### 11.10.3. Deliverables

| Delivery | Description |
|----------|-------------------------------------|
| SAC | Final Statistical Analysis Complete |

<sup>•</sup> Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

# 11.10.4. Study Population Tables

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Subjec | t Disposition | | | | |
| 1.1. | All Treated<br>Subjects | ES1 | Summary of Participant Disposition for the Participant Conclusion Record | ICH E3, FDAAA, EudraCT | SAC |
| 1.2. | All Treated<br>Subjects | SD1 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | | SAC |
| 1.3. | Enrolled | NS1 | Summary of Number of Participant by Country and Site ID | EudraCT/Clinical Operations | SAC |
| Demog | raphic and Base | line Characteristics | | | |
| 1.4. | All Treated<br>Subjects | DM1 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT | SAC |
| 1.5. | Enrolled | DM11 | Summary of Age Ranges | EudraCT | SAC |
| 1.6. | All Treated<br>Subjects | DM5 | Summary of Race and Racial Combinations | ICH E3, FDA, FDAAA, EudraCT | SAC |
| Medica | al History and C | oncomitant Medic | cations | | |
| 1.7. | All Treated<br>Subjects | MH1 | Summary of Current/Past Medical Conditions | | SAC |
| 1.8. | All Treated<br>Subjects | CM8 | Summary of Concomitant Medications | Include both prior and concomitant medications | SAC |
| Exposi | Exposure and Treatment Compliance | | | | |
| 1.9. | All Treated<br>Subjects | POP_T1 | Summary of Exposure to GSK2879552 | Include 2mg QD/ATRA<br>45mg/m2/day | SAC |

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 1.10. | All Treated<br>Subjects | ODMOD1 | Summary of Dose Reductions to GSK2879552 | | SAC |
| 1.11. | All Treated<br>Subjects | ODMOD8 | Summary of Dose Escalations to GSK2879552 | | SAC |
| 1.12. | All Treated<br>Subjects | ODMOD2 | Summary of Dose Interruptions to GSK2879552 | | SAC |
| Prior A | nti-Cancer The | rapy and Surgical | Procedures | | |
| 1.13. | All Treated<br>Subjects | AC1 | Summary of Prior Anti-Cancer Therapy | | SAC |
| 1.14. | All Treated<br>Subjects | AC3 | Summary of Number of Prior Anti-Cancer Therapy Regimens | | SAC |
| 1.15. | All Treated<br>Subjects | OSP1 | Summary of Cancer Related Surgical Procedures | | SAC |

# 11.10.5. Efficacy Tables

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Clinical | Response | | | | |
| 2.1. | All Treated<br>Subjects | Re1a | Summary of Investigator-Assessed Best Response (Without Confirmation) | <ol> <li>Investigator Assessed Responses would be reported. No confirmation on responses are required.</li> <li>Include the response categories collected in eCRF. i.e. 1. Complete remission (CR) 2. As per CR but PLT &lt; 100 x10^9/L (CRp) 3. Morphologic leukaemia- free state(MLFS) 4. Partial remission (PR) 5. Stable disease 6. Progressive Disease or Relapse of Disease 7. Not evaluable</li> <li>Include just the first two segments of the template. i.e. Best Response and Response rate.</li> <li>Response rate = CR+CRp+MLFS+PR</li> <li>P-value for response rate would not be reported.</li> </ol> | SAC |

# 11.10.6. Safety Tables

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Advers | e Events (AEs) | | | | |
| 3.1. | All Treated<br>Subjects | OAE7 | Summary of All Adverse Events by Maximum Grade by System Organ Class and Preferred Term | | SAC |
| 3.2. | All Treated<br>Subjects | AE3 | Summary of All Adverse Events by System Organ Class and Preferred Term | | SAC |
| 3.3. | All Treated<br>Subjects | AE13 | Overview of Adverse Events | | SAC |
| 3.4. | All Treated<br>Subjects | IDSL AE's of<br>Special Interest<br>– EXAMPLE<br>METABOLIC<br>14.1 | Summary of All Adverse Events of Special Interest | | SAC |
| 3.5. | All Treated<br>Subjects | AE15 | Summary of Common (>=5%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Participant and Occurrences) | FDAAA, EudraCT | SAC |
| Serious | Serious and Other Significant Adverse Events | | | | |
| 3.6. | All Treated<br>Subjects | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Participants and Occurrences) | FDAAA, EudraCT | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Pleasel | _aboratory: Ch | emistry | | | |
| 3.7. | All Treated<br>Subjects | OLB9C | Summary of Clinical Chemistry Toxicity Grade Change from Baseline Grade | For gradable Clinical chemistry tests. By dose, and overall. Include Worst-case. | SAC |
| 3.8. | All Treated<br>Subjects | OLB11C | Summary of Clinical Chemistry Laboratory Changes from Baseline with Respect to the Normal Range | For non-gradable lab tests. By dose, and overall. | SAC |
| Labora | tory: Hematolo | gy | | | |
| 3.9. | All Treated<br>Subjects | OLB9C | Summary of Haematology Toxicity Grade Change from Baseline Grade | For gradable Haematology tests. By dose, and overall. Include Worstcase. | SAC |
| 3.10. | All Treated<br>Subjects | OLB11C | Summary of Clinical Hematology Laboratory Changes from Baseline with Respect to the Normal Range | For non-gradable lab tests. By dose, and overall. | SAC |
| Labora | tory: Hepatobil | iary (Liver) | | | |
| 3.11. | All Treated<br>Subjects | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities | | SAC |
| ECG | | | | | |
| 3.12. | All Treated<br>Subjects | EG1 | Summary of ECG Findings | | SAC |
| 3.13. | All Treated<br>Subjects | EG10 | Summary of Maximum QTc Values Post-Baseline Relative to Baseline by Category | | SAC |
| 3.14. | All Treated<br>Subjects | EG11 | Summary of Maximum Increase in QTc Values Post-Baseline Relative to Baseline by Category | | SAC |
| 3.15. | All Treated<br>Subjects | SAF_T1 | Summary of Maximum QTc Grades Post-Baseline Relative to Baseline | | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.16. | All Treated<br>Subjects | SAF_T1 | Summary of Maximum Increase in QTc Grades Post-Baseline Relative to Baseline | | SAC |
| Vital Si | gns | | | | |
| 3.17. | All Treated<br>Subjects | OVT1B | Summary of Changes in Heart Rate from Baseline | | SAC |
| 3.18. | All Treated<br>Subjects | OVT2B | Summary of Increases in Blood Pressure from Baseline | | SAC |
| 3.19. | All Treated<br>Subjects | OVT1B | Summary of Changes in Temperature from Baseline | The following categories need to be included: Decrease to <=35 Change to normal or no change Increase to >=38 | SAC |
| ECOG | | | | | |
| 3.20. | All Treated<br>Subjects | PS4A | Summary of Change in ECOG 'Performance Status' from Baseline | | SAC |

### 11.10.7. Pharmacokinetic Tables

| Pharm | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| PK Co | ncentration | | | | |
| 4.1. | 4.1. Pharmacokinetic PK01 Summary of GSK2879552 Plasma Pharmacokinetic Concentration-Time Data | | | SAC | |
| PK Pa | rameters | | | | |
| 4.2. | Pharmacokinetic | PK06 | Summary of Derived GSK2879552 Plasma Pharmacokinetic Parameters (non-transformed and log-transformed) | | SAC |
| 4.3. | Pharmacokinetic | PK_T1 | Summary of Statistical Analysis to Assess the Dose<br>Proportionality for AUC (0-∞) and Cmax Using Power Model –<br>Day 1 | | SAC |
| 4.4. | Pharmacokinetic | PK_T1 | Summary of Statistical Analysis to Assess the Dose<br>Proportionality for AUC (0- z) and Cmax Using Power Model –<br>Day 15 | | SAC |
| 4.5. | Pharmacokinetic | PK_T2 | Summary of Statistical Analysis to Assess the Accumulation for AUC $(0-\tau)$ on Day 15 vs AUC $(0-\tau)$ on Day 1 by Dose | | SAC |
| 4.6. | Pharmacokinetic | PK_T2 | Summary of Statistical Analysis to Assess the Time Invariance based on AUC(0- $\infty$ ) on Day 1 and AUC(0- $\tau$ ) on Day 15 by Dose | | SAC |

# 11.10.8. ICH Listings

| ICH: Li | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Subjec | t Disposition | | | | |
| 1. | Screened | ES7 | Listing of Reasons for Screen Failure | Journal Guidelines | SAC |
| 2. | All Treated<br>Subjects | ES2 | Listing of Reasons for Study Withdrawal | | SAC |
| 3. | All Treated<br>Subjects | SD2 | Listing of Reasons for Study Treatment Discontinuation | Remove "Number of cycles" column. Add investigational product as one of the column | SAC |
| Protoc | ol Deviations | | | | |
| 4. | All Treated<br>Subjects | DV2 | Listing of Important Protocol Deviations | | SAC |
| 5. | Screened | IE3 | Listing of Participants with Inclusion/Exclusion Criteria Deviations | | SAC |
| Popula | ations Analysed | | | | |
| 6. | Enrolled | SP3 | Listing of Participants Excluded from Any Population | | SAC |
| Demog | graphic and Bas | eline Characteris | tics | | |
| 7. | All Treated<br>Subjects | DM2 | Listing of Demographic Characteristics | | SAC |
| 8. | All Treated<br>Subjects | DM9 | Listing of Race | | SAC |
| Medica | al History and C | oncomitant Medic | cations | | |
| 9. | All Treated<br>Subjects | MH2 | Listing of Past/Current Medical Conditions | Oncology specific template to be used | SAC |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 10. | All Treated<br>Subjects | OCM1A | Listing of Concomitant Medications | Include both prior and concomitant medications | SAC |
| Exposi | ure and Treatmo | ent Compliance | | | |
| 11. | All Treated<br>Subjects | EX3 | Listing of Exposure Data | Include a flag variable to indicate imputed date. | SAC |
| 12. | All Treated<br>Subjects | ODMOD10A | Listing of Dose Reductions | | SAC |
| 13. | All Treated<br>Subjects | ODMOD11A | Listing of Dose Interruptions | | SAC |
| 14. | All Treated<br>Subjects | ODMOD15A | Listing of Dose Escalations | | SAC |
| Advers | e Events | | | | |
| 15. | All Treated<br>Subjects | OAE04 | Listing of All Adverse Events | | SAC |
| 16. | All Treated<br>Subjects | OAE03 | Listing of Subject Numbers for Individual Adverse Events | | SAC |
| 17. | All Treated<br>Subjects | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | | SAC |
| 18. | All Treated<br>Subjects | OAE04 | Listing of Encephalopathy: Adverse Event of Special Interest | | SAC |
| 19. | All Treated<br>Subjects | OAE04 | Listing of Thrombocytopenia: Adverse Event of Special Interest | | SAC |
| 20. | All Treated<br>Subjects | OAE04 | Listing of Hemorrhages: Adverse Event of Special Interest | | SAC |

| ICH: Lis | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 21. | All Treated<br>Subjects | OAE04 | Listing of Diarrhoea: Adverse Event of Special Interest | | SAC |
| 22. | All Treated<br>Subjects | OAE04 | Listing of Nausea and Vomiting: Adverse Event of Special Interest | | SAC |
| 23. | All Treated<br>Subjects | OAE04 | Listing of Constipation: Adverse Event of Special Interest | | SAC |
| 24. | All Treated<br>Subjects | OAE04 | Listing of Infections: Adverse Event of Special Interest | | SAC |
| 25. | All Treated<br>Subjects | OAE04 | Listing of Neutropenia: Adverse Event of Special Interest | | SAC |
| 26. | All Treated<br>Subjects | OAE04 | Listing of Fatigue: Adverse Event of Special Interest | | SAC |
| 27. | All Treated<br>Subjects | OAE04 | Listing of Anaemia: Adverse Event of Special Interest | | SAC |
| Serious | and Other Signific | ant Adverse Events | | | |
| 28. | All Treated<br>Subjects | OAE4 | Listing of Fatal Serious Adverse Events | | SAC |
| 29. | All Treated<br>Subjects | OAE4 | Listing of Non-Fatal Serious Adverse Events | | SAC |
| All Lab | oratory | | | | |
| 30. | All Treated<br>Subjects | OLB7 | Listing of Clinical Chemistry Laboratory Data | | SAC |
| 31. | All Treated<br>Subjects | OLB7 | Listing of Haematology Laboratory Data | | SAC |

| ICH: Listings | | | | |
|---|---|---|---|---|
| No. | o. Population IDSL / Example Shell Title Programming Notes | | | |
| ECG | | | | |
| 32. | All Treated<br>Subjects | EG3 | Listing of ECG Values | SAC |
| 33. | All Treated<br>Subjects | EG5 | Listing of Abnormal ECG Findings | SAC |
| Vital Sig | Vital Signs | | | |
| 34. | All Treated<br>Subjects | VS4 | Listing of Vital Signs | SAC |

# 11.10.9. Non-ICH Listings

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| Substa | Substance Use | | | | |
| 35. | All Treated Subjects | SU2 | Listing of Substance Use | | SAC |
| Prior A | anti-Cancer Therapy an | d Surgical P | rocedure | | |
| 36. | All Treated Subjects | AC6 | Listing of Prior Anti-Cancer Therapy Regimens | | SAC |
| 37. | All Treated Subjects | OSP3 | Listing of Cancer Related Surgical Procedures | | SAC |
| Blood | Products | | | 1 | |
| 38. | All Treated Subjects | BP4 | Listing of Blood Products | | SAC |
| Diseas | e Characteristics | | | | |
| 39. | All Treated Subjects | POP_L1 | Listing of Disease Characteristics at Screening | | SAC |
| Efficac | sy . | | | | |
| 40. | All Treated Subjects | EFF_L1 | Listing of Investigator-Assessed Responses (Without Confirmation) | | SAC |
| Safety | | | | | |
| 41. | All Treated Subjects | OLVEF2A | Listing of Left Ventricular Ejection Fraction Results | | SAC |
| 42. | All Treated Subjects | PS5A | Listing of ECOG Performance Status | | SAC |
| 43. | All Treated Subjects | SAF_L1 | Listing of Montreal Cognitive Assessment (MOCA) | | SAC |
| 44. | All Treated Subjects | DTH3 | Listing of Death | | SAC |
| 45. | All Treated Subjects | LIVER6 | Listing of Liver Stopping Event Information for RUCAM Score | | SAC |

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| PK | | | | | |
| 46. | Pharmacokinetic | PK07 | Listing of GSK2879552 Plasma PK Concentration-Time Data | | SAC |
| 47. | Pharmacokinetic | PK07 | Listing of ATRA Plasma PK Concentration-Time Data | | SAC |
| 48. | Pharmacokinetic | PK13 | Listing of GSK2879552 Plasma PK Parameters Data | | SAC |

## 11.11. Appendix 11: Example Mock Shells for Data Displays

Example: POP\_T1 Page 1 of n

Protocol: 200200

Population: All Treated Subjects

# Table X Summary of Exposure to GSK2879552

| | | 1mg QD | 2mg QD | 4mg QD | 8mg QD | 12mg QD | 20mg QD |
|---|---|---|---|---|---|---|---|
| Duration of Exposure(weeks) [1] | n | X | X | X | X | X | X |
| | Mean | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX |
| | SD | X.XXXX | X.XXXX | X.XXXX | X.XXXX | X.XXXX | X.XXXX |
| | Median | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX |
| | Min. | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Max. | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| Average Daily<br>Dose(mg) [2] | n | X | X | X | X | X | X |
| | Mean | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX |
| | SD | X.XXXX | X.XXXX | X.XXXX | X.XXXX | X.XXXX | X.XXXX |

200200

| Median | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX |
|--------|-------|-------|-------|-------|-------|-------|
| Min. | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |
| Max. | X.XX | X.XX | X.XX | X.XX | X.XX | X.XX |

Note: [1] Duration of exposure = end date of GSK2879552 - start date of GSK2879552 + 1.

<sup>[2]</sup> Average daily dose = Cumulative dose divided by duration of exposure.

200200

Example: POP\_L1 Protocol: 200200 Page 1 of n

Population: All Treated Subjects

## Listing X

## Listing of Disease Characteristics at Screening

Treatment: 1mg QD

| Centre<br>Id/<br>Subj. | Visceral or non-<br>visceral disease | Date of Last<br>Recurrence/Time<br>since<br>recurrence(days) | Date of Last<br>Progression/Time<br>since<br>progression(days) | WHO classification<br>of AML/WHO<br>classification of<br>AML subtype | FAB<br>classification<br>of AML | Lines of<br>therapy<br>completed<br>Screen | History<br>of<br>CNS<br>lesions |
|---|---|---|---|---|---|---|---|
| PPD | Non-visceral | 25AUG2014/<br>64 | 25AUG2014/<br>64 | AML, not otherwise categorized/AML with maturation | M2 | 4 lines | N |

200200

Example: EFF\_L1 Page 1 of n

Protocol: 200200

Population: All Treated Subjects

# Listing X Listing of Investigator-Assessed Responses (Without Confirmation)

Treatment: 1mg QD

| Centre Id/ | Age(y)/ | Visit | Date | Resp. Day | Response Assessment |
|---|---|---|---|---|---|
| Subj. | Sex/ | | | | |
| | Race | | | | |
| PPD | 68/ | Day 15 | PPD | 16 | Stable disease |
| | M/ | | | | |
| | White - | | | | |
| | White/Caucasian/European | | | | |
| | Heritage | | | | |

Example: SAF\_T1 Protocol: 200200 Page 1 of n

Population: All Treated Subjects

Table X
Summary of Maximum QTc Grades Post-Baseline Relative to Baseline

| | | | Corrected QT (Friedericia's correction) interval (MSEC) | | | | | |
|---|---|---|---|---|---|---|---|---|
| Treatment | N | interval (MSEC) | | | | Grade 2 | Grade 3 | Missing |
| 1mg QD | 1 | Grade 0<br>Grade 1<br>Grade 2<br>Grade 3<br>Missing | 0 | | 0<br>0<br>0 | | 0<br>0<br>0<br>0 | 0<br>0<br>0<br>0 |
| 2mg QD | 2 | Grade 0<br>Grade 1<br>Grade 2<br>Grade 3<br>Missing | 1<br>0<br>0 | (50%)<br>(50%) | 0<br>0<br>0 | 0<br>0<br>0<br>0 | 0<br>0<br>0<br>0 | 0<br>0<br>0<br>0 |
| 4mg QD | 7 | Grade 0<br>Grade 1<br>Grade 2<br>Grade 3<br>Missing | 0 | | 0<br>0 | 0<br>0<br>0<br>0 | 0<br>0<br>0<br>0 | 0<br>0<br>0<br>0 |
| 8mg QD | 5 | Grade 0<br>Grade 1<br>Grade 2<br>Grade 3<br>Missing | 1<br>0<br>0 | (33%)<br>(33%)<br>(33%) | 0<br>0<br>0 | 0<br>0<br>0<br>0 | 0<br>0<br>0<br>0 | 0<br>0<br>0<br>0 |

200200

Example: SAF\_L1 Page 1 of n
Protocol: 200200

Population: All Treated Subjects

# Listing X Listing of Montreal Cognitive Assessment (MOCA)

| Treatment | Centre | Age(y)/ | Visit | Date of | MOCA | MOCA |
|---|---|---|---|---|---|---|
| | ID/ | Sex/ | | Assessment/Time | Education | Total Score |
| | Subj. | Race | | of Assessment | | |
| | | | | Study day | | |
| 8.0mg QD | PPD | 68/ | SCREENING | PPD | <= 12 years | 26 |
| | | M/ | | 10:30 | education | |
| | | White - | | -4 | | |
| | | White/Caucasian/European | | | | |
| | | Heritage | | | | |

200200

Example: PK\_T1 Page 1 of n

Protocol: 200200

Population: Pharmacokinetic

Table X Summary of Statistical Analysis to Assess the Dose Proportionality for  $AUC(0-\infty)$  and Cmax Using Power Model – Day 1

| | | | 90% Confidence Interval | |
|---|---|---|---|---|
| Parameter | Number of subjects | Estimated Mean Slope | 90% CI Low | 90% CI High |
| AUC(0-inf) | XX | X.XXX | X.XXX | X.XXX |
| Cmax | XX | X.XXX | X.XXX | X.XXX |

Note: Repeat the same for Table No. 4.5: Summary of Statistical Analysis to Assess the Dose Proportionality for  $AUC(0-\tau)$  and Cmax Using Power Model – Day 15

200200

Example: PK\_T2 Page 1 of n

Protocol: 200200

Population: Pharmacokinetic

Table X Summary of Statistical Analysis to Assess the Accumulation for AUC  $(0-\tau)$  on Day 15 vs AUC $(0-\tau)$  on Day 1 by Dose

| Treatment | | Geometric LSMean | | Comparison | | 90% Confidence |
|---|---|---|---|---|---|---|
| | n | Test | Ref. | Test/Ref. | Ratio | Interval |
| 1mg QD | X | XX.XX | XX.XX | Day 15 vs Day 1 | X.XXX | (X.XXX, X.XXX) |
| 2mg QD | X | XX.XX | XX.XX | Day 15 vs Day 1 | X.XXX | (X.XXX, X.XXX) |

Note: Repeat the same for Table No. 4.7: Summary of Statistical Analysis to Assess the Time Invariance based on  $AUC(0-\infty)$  on Day 15 by Dose